CLINICAL TRIAL: NCT00306020
Title: Analgesia and Wound Healing Assessment Following Topical Morphine Applied to Patients With Cutaneous Cancer Related Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn due to difficulties in recruiting appropriate patients in community clinic setting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Israel Cancer Association (Other)
Responsible Party: Principal Investigator, Pesach Shvartzman, Head-Department of Family Medicine, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOR394105CTIL
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Ulcer; Wounds and Injuries
Keywords: Skin ulcers; Topical morphine; Chronic pain; Cancer
MeSH Terms: conditions — Ulcer; Wounds and Injuries; Skin Ulcer; Chronic Pain; Neoplasms | interventions — Morphine

INTERVENTIONS:
Drug: topical morphine

SUMMARY:
Cutaneous cancer-related pain is difficult to treat. These patients are often prescribed high systemic dosages of opioids. Yet, many patients continue to report pain while experiencing dose-limiting side effects. An alternative approach to systemic administration is to apply topical medications. The advantage of topical application is the potential of achieving good analgesia using low dosages with few, if any, systemic side effects. Current clinical data indicates, that topically applied morphine has an analgesic effect in patients with severe pain and that it may even improve wound healing. The clinical reports so far have been either case studies or double blind randomly controlled trials with a very small sample size of patients. There is still a great deal of information which is lacking about this modality of treatment regarding on the one hand, the mechanism of action and on the other, clinical issues. For example, is the mechanism of the effect actually peripheral? What is the adequate dose of analgesic medication for different types of skin conditions? Wound healing has not been quantified.

We will apply morphine topically to skin wounds of cancer and evaluate the effect of the treatment on pain, side effects, quantify wound healing, quantify morphine and its metabolites in blood and urine.

Should well controlled studies, demonstrate all or any of the peripheral effects of topical morphine, clinical application of this treatment modality would be possible. This could contribute towards better treatment of these patients, who have pain which is difficult to treat and can, at times, be intractable.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe resting pain (scores above 5/10).
* Stable analgesic regimen.
* No surgical interventions planned during the study period.
* Able to self-assess pain and report it.
* Hospitalized or receiving home care for Stage I; out-patients or receiving home care for Stage II.
* Wound not infected or covered with necrotic tissue.

Exclusion Criteria:

* True sensitivity to opioids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pain intensity reports
frequency and type of side effects
blood and urine levels of morphine and its metabolites, morphine 3- and 6-glucuronide

SECONDARY OUTCOMES:
quantification of wound healing
change in use of regular analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Shvartzman, Professor, Principal Investigator — Ben-Gurion University of the Negev, Sial Research Center for Family Medicine and Primary Care